CLINICAL TRIAL: NCT05633784
Title: Telemedicine Home-based Management in Patients With Chronic Heart Failure and Type 2 Diabetes: a Randomized Control Study
Brief Title: Telemedicine Home-based Management in Patients With CHF and Type 2 Diabetes
Acronym: TELEMECHRON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Azienda Ospedaliera Bolognini di Seriate Bergamo (Other); Papa Giovanni XXIII Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICS Maugeri CE2338; NET-2018-12367206-WP3 (Other: Italian Ministry of Health)
Record Dates: First submitted 2022-11-17; First posted 2022-12-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Chronic Heart Failure; Diabetes Mellitus
Keywords: telemedicine; case management; mobile technologies (mHealth); Physical activities; 6-min walking test; motivational feedback
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity | interventions — Remote Consultation; Telerehabilitation; Telemedicine; Quality of Life

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Consenting eligible patients were randomized to either an Intervention or a Control group (1:1).
  A computer (www.randomization.com) generated tables to allocate patients in fixed blocks of four. In order to prevent selection bias, the list of randomization will be managed by personnel not directly involved in the enrolment of the patient. Due to the nature of the intervention, neither the patients nor the physicians were blinded to patients' group allocation. However, outcome assessors and data analysts will be blinded to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): At the beginning and at the end of the 6-month study period, patients of the Intervention group will perform outpatient cardiological visits. During the 6-month they will be followed through a home remote teleassistance program, designed to provide multidisciplinary support.
  Interventions: Other: Teleassistance; Other: Teleconsultation; Other: Telerehabilitation; Other: Telemonitoring; Other: mHealth; Other: telepsycology; Other: Quality of life; Other: Biochemistry evaluation; Other: Clinical evaluation; Other: State of health of the patient
- Control group (Active Comparator): At the beginning and at the end of the 6-month study period, patients of the Control group will perform outpatient cardiological visits. During the 6-month at home, patients will be followed in the usual care model by GP.
  Interventions: Other: Quality of life; Other: Biochemistry evaluation; Other: Clinical evaluation; Other: State of health of the patient

INTERVENTIONS:
Other: Teleassistance — Support the nursing case manager through a structured teleconsultation program (telephone and videoconference support at least once a week)
  Arms: Intervention group
Other: Teleconsultation — Cardiological and Diabetological teleconsultation at the beginning of the program and in case of need during the program.
  Arms: Intervention group
Other: Telerehabilitation — Support from a physiotherapist (if needed)
  Arms: Intervention group
Other: Telemonitoring — Telemonitoring of patient vital signs (eg single electrocardiographic trace) and delay steps
  Arms: Intervention group
Other: mHealth — The support of an App for recording and monitoring parameters: delay treatment, clinical parameters such as glycemia, blood pressure, HR, symptoms, etc.
  Arms: Intervention group
Other: telepsycology — Psychological support (if necessary)
  Arms: Intervention group
Other: Quality of life — Minnesota LIVING WITH HEART FAILURE® Questionnaire (MLHFQ), Short Form Survey (SF-12) Questionnaire and Diabetes Quality of Life (DQoL) questionnaire
Other: Biochemistry evaluation — Glycemia, glycated haemoglobin, total cholesterol, HDL and LDL, triglycerides, creatinine, BUN, creatinine clearance, BNP
Other: Clinical evaluation — 6-minute-walking test, IMC, NYHA class, Ejection fraction
Other: State of health of the patient — Severity Index and Comordbidity index

SUMMARY:
The progressive ageing of the population of industrialized countries is accompanied by a dramatic increase in the prevalence of chronic multi-pathologies. In the general population, HF is associated with a higher prevalence of T2DM compared with patients without HF and with marked regional differences observed in Europe and the rest of the world. In clinical trials of chronic HF patients, the prevalence of T2DM is approximately 30% in patients with reduced or preserved ejection fraction and rises to as much as 45% in hospitalized patient registries. A complex drug regimen is often associated with low adherence in patients with HF and T2DM and poor adherence is associated with adverse clinical events. Similarly, adherence to recommendations regarding lifestyle changes, such as increasing physical activity, is often limited despite these changes' favourable effects on the patient. Therefore, interventions are needed to improve all these factors and optimize adherence. The inclusion of telemedicine (telenursing, telerehabilitation, mHealth) focused on health and correct behaviour can create opportunities to implement customized and scalable solutions in populations at risk. The project will aim to evaluate for patients with chronic diseases with a complex phenotype (heart failure and type II diabetes mellitus) the effectiveness of a remote surveillance program with particular attention to lifestyle changes.

ELIGIBILITY:
Inclusion Criteria:

* Inform consent
* Age ≥ 18 years
* Documented diagnosis of heart failure, NYHA class II-III (reduced or preserved Ejection fraction without hospitalization in the last 3 months
* Diagnosis of Diabetes Mellitus Type II in pharmacological treatment from at least one month
* Ability to walk without assistive devices
* Consent to using a device (independently or with the support of a caregiver) for recording the single electrocardiographic trace at home
* Consent to using the App

Exclusion Criteria:

* Subjects with poor collaboration
* No possibility of using mobile technology
* Life expectancy of fewer than 6 months
* Medical issues that preclude participation in the program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in tolerance capacity | Baseline and 6 months
  The change from baseline in tolerance capacity will be measured by walking test performance (meters walked).

SECONDARY OUTCOMES:
Change of hospitalizations | 6 months
  Change of hospitalizations for cardiovascular problems, diabetes and all-causes
Number of Steps | Baseline and 6 months
  The difference in the weekly mean in the number of steps from baseline over the 6 months of follow-up.
HbA1c dosage | Baseline and 6 months
  Change of the disease status
Change in quality of life related to heart failure | Baseline and 6 months
  Change in quality of life measured by Minnesota Living with Heart Failure (MLHFQ) questionnaire
Change in quality of life related to Diabetes | Baseline and 6 months
  Change in quality of life measured by Diabetes quality of life (DQoL) questionnaire
Change in quality of life | Baseline and 6 months
  Change in quality of life measured by 12-item Short Form Survey (SF-12) questionnaire
Assessment of physical activity. | Baseline and 6 months
  Change in physical activity profile by Physical Activity Scale for the Elderly (PASE).
  The total PASE score is computed by multiplying the amount of time spent on each activity (hours/week) or participation (yes/no) in an activity by the empirically derived item weights and summing overall activities.

CONTACTS AND LOCATIONS:
Overall Officials: SIMONETTA SCALVINI, MD, Study Chair — ICS MAUGERI
Locations (3):
- Italy (3):
  - Azienda Ospedaliera Bolognini di Seriate Bergamo, Seriate, Bergamo
  - Istituti Clinici Scientifici Maugeri, Lumezzane, Brescia
  - Papa Giovanni XXIII Hospital, Bergamo

REFERENCES:
- [Background] Seferovic PM, Petrie MC, Filippatos GS, Anker SD, Rosano G, Bauersachs J, Paulus WJ, Komajda M, Cosentino F, de Boer RA, Farmakis D, Doehner W, Lambrinou E, Lopatin Y, Piepoli MF, Theodorakis MJ, Wiggers H, Lekakis J, Mebazaa A, Mamas MA, Tschope C, Hoes AW, Seferovic JP, Logue J, McDonagh T, Riley JP, Milinkovic I, Polovina M, van Veldhuisen DJ, Lainscak M, Maggioni AP, Ruschitzka F, McMurray JJV. Type 2 diabetes mellitus and heart failure: a position statement from the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2018 May;20(5):853-872. doi: 10.1002/ejhf.1170. Epub 2018 Mar 8. PMID 29520964
- [Background] Thrainsdottir IS, Aspelund T, Thorgeirsson G, Gudnason V, Hardarson T, Malmberg K, Sigurdsson G, Ryden L. The association between glucose abnormalities and heart failure in the population-based Reykjavik study. Diabetes Care. 2005 Mar;28(3):612-6. doi: 10.2337/diacare.28.3.612. PMID 15735197
- [Background] Sharma A, Mentz RJ, Granger BB, Heitner JF, Cooper LB, Banerjee D, Green CL, Majumdar MD, Eapen Z, Hudson L, Felker GM. Utilizing mobile technologies to improve physical activity and medication adherence in patients with heart failure and diabetes mellitus: Rationale and design of the TARGET-HF-DM Trial. Am Heart J. 2019 May;211:22-33. doi: 10.1016/j.ahj.2019.01.007. Epub 2019 Jan 31. PMID 30831331
- [Background] Scalvini S, Bernocchi P, Zanelli E, Comini L, Vitacca M; Maugeri Centre for Telehealth and Telecare (MCTT). Maugeri Centre for Telehealth and Telecare: A real-life integrated experience in chronic patients. J Telemed Telecare. 2018 Aug;24(7):500-507. doi: 10.1177/1357633X17710827. Epub 2017 May 24. PMID 28537509
- [Background] Bernocchi P, Giudici V, Borghi G, Bertolaia P, D'Isa S, Trevisan R, Scalvini S. Telemedicine home-based management in patients with chronic heart failure and diabetes type II: study protocol for a randomized controlled trial. Trials. 2024 May 21;25(1):333. doi: 10.1186/s13063-024-08171-0. PMID 38773662